CLINICAL TRIAL: NCT06501716
Title: I See G: Superior Hypophyseal Artery Intraoperative Indocyanine Green Angiogram as a Predictor of Postoperative Visual Function After Endoscopic Endonasal Surgery
Brief Title: ICG Angiogram as a Predictor of Postoperative Visual Function After EEA Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 24-41191
Record Dates: First submitted 2024-06-30; First posted 2024-07-15 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Indocyanine Green; Skull Base Neoplasms
MeSH Terms: conditions — Skull Base Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICG Group: Eligible participants are those diagnosed with suprasellar lesions undergoing ICG angiography during endoscopic endonasal resection.
  Interventions: Procedure: Indocyanine Green

INTERVENTIONS:
Procedure: Indocyanine Green — Tumor resection, direct visualization of the chiasm and both optic nerves and ICG administration will be provided as it is recommended by the standard of care. ICG will be administered by an injection of 5 mg of ICG diluted in a 10 mL syringe performed in the line closest to the heart followed by a 10-mL saline bolus. Using near-infrared lighting, the investigators will determine the time between anterior cerebral arteries (ACA) peak luminescence to the peak luminescence of the superior hypophyseal arteries enveloping the optic chiasm (ACA to chiasm time). Because luminescence of large vessels precedes small arterial penetration, signal from the ACAs was considered as "time 0" to account for possible differences in the arm-brain time between patients. In addition, the investigators will analyze the proportion of superior hypophyseal branches on the chiasm that luminesced from ICG.

SUMMARY:
Endonasal endoscopic approaches are an established treatment for suprasellar lesions compromising the optic nerves (ON). Surgery often involves dissecting tumors from the optic nerves and its blood supply, which can result in nerve damage and visual loss after surgery. To date, there are no reliable methods to monitor the optic nerve function during surgery and thus, post-surgical visual outcomes is unknown until the patients are fully awake after surgery for a visual exam. This delay in diagnosis prevents early therapeutic measures and can result in further harm to the ON. We have recently recognized that when ICG is routinely injected during these cases to check for patency of the big arteries the sub millimetric superior hypophyseal arteries supplying (SHA) the ON are also visible and that lack of visualization of these vessels is associated with worse visual deficits after surgery. Thus, ICG may be a tool to intraoperative predict visual outcomes after endonasal approach for suprasellar lesions and fill the nondiagnostic gap. This study will assess whether endoscopic ICG angiography before and after resection of suprasellar lesions can predict post-operative visual deficits. Successful completion will provide surgeons a novel tool to assess visual function during surgery. The ICG endoscopic angiograms suggested in this study are noninvasive and currently routinely performed at the end of surgery to check for patency of big brain arteries.

ELIGIBILITY:
Inclusion Criteria:

* The study will enroll adult (18 y.o. and older) participants undergoing endonasal endoscopic surgery for suprasellar tumors including meningiomas, craniopharyngiomas and pituitary adenomas.

Exclusion Criteria:

* Underage patients (younger than 18 y.o).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed in the clinic with sellar or suprasellar pituitary tumors and scheduled for an endoscopic endonasal surgical resection will be approached to obtain consent to participate in this study. These patients will be identified by the PI of this study who will recommended the use of ICG based in the tumor characteristics and risk-benefit potential for the patient.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with Post Operative Visual Acuity Impairment and Visual Field Defect | From the surgery to first post-operative follow up (6 weeks)
  The investigators will evaluate the percentage of participants that present with decreased of visual acuity and any modality of visual field defect after the surgery. Postoperative visual acuity and visual field testing will be performed at 6 weeks postoperative follow up visit to evaluate chiasm function, including cranial nerve examination, bilateral number counting, letter reading, and number identification in 4 quadrants of peripheral vision. Visual evaluations will be performed by the ophthalmology service following our standard postoperative protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Goldschmidt, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osorio RC, Aabedi AA, El-Sayed IH, Gurrola J 2nd, Goldschmidt E. Superior Hypophyseal Artery Intraoperative Indocyanine Green Angiogram as a Predictor of Postoperative Visual Function After Endoscopic Endonasal Surgery. Oper Neurosurg. 2023 Oct 1;25(4):379-385. doi: 10.1227/ons.0000000000000809. Epub 2023 Jun 27. PMID 37366631
- [Background] Shahein M, Prevedello DM, Beaumont TL, Ismail K, Nouby R, Palettas M, Prevedello LM, Otto BA, Carrau RL. The role of indocyanine green fluorescence in endoscopic endonasal skull base surgery and its imaging correlations. J Neurosurg. 2020 Nov 13;135(3):923-933. doi: 10.3171/2020.6.JNS192775. Print 2021 Sep 1. PMID 33186906
- [Background] Ramesh R, Gurrola JG 2nd, Goldschmidt E. Use of Real-Time Superior Hypophyseal Artery Indocyanine Green Angiogram During Endoscopic Resection of a Third Ventricular Craniopharyngioma: 2-Dimensional Operative Video. Oper Neurosurg. 2025 Jan 1;28(1):123-124. doi: 10.1227/ons.0000000000001225. Epub 2024 Jun 7. No abstract available. PMID 38847508
- [Background] Lee MH, Lee TK. Application of fusion-fluorescence imaging using indocyanine green in endoscopic endonasal surgery. J Clin Neurosci. 2022 Apr;98:45-52. doi: 10.1016/j.jocn.2022.01.023. Epub 2022 Feb 4. PMID 35131724